CLINICAL TRIAL: NCT01578798
Title: Detection of Immune Changes as a Result of Surgical Trauma in Human Subject
Status: Completed | Type: Observational
Sponsor: Martin Angst (Other)
Responsible Party: Sponsor-Investigator, Martin Angst, Professor of Anesthesia, Stanford University
Organization: Stanford University (Other)
Other Study IDs: 22678
Record Dates: First submitted 2012-03-23; First posted 2012-04-17 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Surgical Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Surgical trauma triggers a massive inflammatory response. Over time, both the innate and adaptive branches of the immune system are affected by surgical trauma. The purpose of this study to characterize the cellular and molecular mechanisms immune response to surgical trauma. Additionally, detailed information about patients' recovery profile will be recorded over a period of 6 weeks, with the eventual goal of linking immune responses to recovery profiles.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 90
* Planning to undergo hip surgery
* Fluent in English
* Willing and able to sign informed consent and HIPAA authorization

Exclusion Criteria:

* Any systemic disease that might compromise the immune system
* Diagnosis of cancer within the last 5 years
* Psychiatric, immunological, and neurological conditions that would interfere with the collection and interpretation of study data
* Pregnancy
* Any other conditions that, in the opinion of the investigators, may compromise a participant's safety or the integrity of the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary hip replacement.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Mass cytometry of immune signaling events | Blood samples for mass cytometry will be drawn at baseline, 1 hour post-op, 24 hours post-op, 3 days post-op, and 6 weeks post-op.
  The primary molecular outcome is the fold change in phosphorylation of signaling proteins.

SECONDARY OUTCOMES:
Surgical Recovery Scale (SRS) | Data will be collected at baseline, daily through the hospitalization, and every 3 days for 6 weeks.
  The surgical recovery scale is a validated questionnaire yielding a numerical score and assessing postoperative recovery.
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Data will be collected at baseline, daily through the hospitalization, and every 3 days for 6 weeks.
  Western Ontario and McMaster Universities Arthritis Index is a validated questionnaires yielding a numerical score and assessing functional status and pain in patients suffering from osteoarthritis of the hip.
Plasma cytokines | Blood samples will be drawn at baseline, 1 hour post-op, 24 hours post-op, 3 days post-op, and 6 weeks post-op.
  The plasma concentration of plasma cytokines and chemokines will be measured with aid of a large protein array.

CONTACTS AND LOCATIONS:
Overall Officials: Martin S Angst, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Hospital, Stanford, California, United States

REFERENCES:
- [Derived] Gaudilliere B, Fragiadakis GK, Bruggner RV, Nicolau M, Finck R, Tingle M, Silva J, Ganio EA, Yeh CG, Maloney WJ, Huddleston JI, Goodman SB, Davis MM, Bendall SC, Fantl WJ, Angst MS, Nolan GP. Clinical recovery from surgery correlates with single-cell immune signatures. Sci Transl Med. 2014 Sep 24;6(255):255ra131. doi: 10.1126/scitranslmed.3009701. PMID 25253674